CLINICAL TRIAL: NCT02756195
Title: The Impact of Non-Routine Events on Neonatal Safety in the Perioperative Environment
Brief Title: The Impact of Non-Routine Events on Neonatal Safety
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Utah (Other)
Responsible Party: Principal Investigator, Dan France, Research Professor of Anesthesiology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 050488; 1R01HD086792-01 (NIH)
Record Dates: First submitted 2016-04-21; First posted 2016-04-29 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Neonatology
Keywords: Patient safety; adverse events; pediatric surgery; quality improvement; health systems; observational study; non-routine event; National Surgical Improvement Program

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Neonates receiving first-time non-cardiac surgery: No intervention will be administered. This is a prospective observational patient safety study focusing on the safety of care delivered to neonates in perioperative care settings. Neonates who receive NICU care both pre- and post-operatively will be eligible for this study.

SUMMARY:
The study objective is to decrease neonatal mortality and morbidity by elucidating the etiology of system failures during perioperative care.

In Aim 1 the investigators will use a novel event discovery method, based on the construct of the nonroutine event (NRE), to efficiently capture dysfunctional clinical microsystem attributes and potentially dangerous conditions. A NRE is defined as any event that is perceived by care providers or skilled observers as a deviation from optimal care based on the clinical situation.

In Aim 2, the investigators will perform a comparative analysis of prospectively collected NRE data to the data collected by conventional event reporting methodologies.

In Aim 3 the investigators will collaborate with Primary Children's Hospital (PCH) in Salt Lake City, UT to conduct practical pilot testing of tools and measures developed and refined in the first two Aims.

Products from Aims 1 & 2 will include:

1. a taxonomy of NREs and outcomes for perioperative neonates;
2. neonatal Comprehensive Open-Ended Non-routine Event Survey (NCONES) data collection tool;
3. comparisons of 5 established event reporting systems, including their rates, costs and benefits; and
4. a guide to prototype neonatal safety surveillance and risk prediction for hospitals and NICUs.

Aim 3 will capitalize on PCH's robust network of NICUs, neonatologists, and patient-level outcome data to conduct a pilot implementation evaluation of the methods and tools developed and refined in Aims 1-2.

DETAILED DESCRIPTION:
Neonates are highly vulnerable to iatrogenic events due to their size, fragility, and severe sensitivity to environmental stressors. Patient safety research in neonatal intensive care units (NICU) has shown that these attributes increase care complexity and reduce the capacity of the neonates to endure even small care deviations. As a result, neonates experience adverse events at rates as high as 8 times of those reported for hospitalized adults. Adverse events are estimated to occur at a rate of 74 events per every 100 NICU patients (0-11 Adverse Event(AE)/patient), with a third being severe events. The vulnerabilities of neonates are most exposed in the perioperative environment, in which little patient safety research has been conducted. In addition to the prevailing risks to all surgical patients (e.g., misidentification, positioning errors, wrong site or side, retained foreign bodies, etc.), neonates are at increased risk to handover (e.g., NICU nurse to Operating Room team), transport (e.g., monitoring), and intraoperative events (e.g., weight-based dosing, temperature control, etc.).

The objective of this multi-site study is to improve neonatal safety by applying a novel event discovery methodology to determine the etiology of system failures in the perioperative environment. The investigators will use the construct of the non-routine event (NRE) to more efficiently capture dysfunctional clinical microsystem attributes and potentially dangerous conditions. A NRE is defined as any event that is perceived by care providers or skilled observers as a deviation from optimal care based on the clinical situation. NREs encompass a substantially larger class of events than conventional patient safety metrics, including sentinel events, medical errors, or "near misses". In prior studies, minimizing the number of deviations from standard care, minor problems, and disruptions during a case has been shown to result in smoother, safer, and shorter surgeries. Moreover, in preliminary studies by members of the research team, intraoperative NREs appeared to be associated with 30-day surgical mortality and morbidity. The Investigators propose a comprehensive 4-year study of neonatal patient safety in the perioperative environment to produce the knowledge base required to inform high-impact intervention studies and guide rapid cycle quality improvement.

The study's Aims are to:

1a) Determine the prevalence and characteristics of NREs during the perioperative care of neonates;

1b) Delineate the relationship(s) between NREs, contributory factors, and surgical mortality and major morbidity during neonatal perioperative care;

2) Perform a comparative analysis of prospective NRE data collection with conventional event reporting methodologies within the same clinical environment; and

3) Collaborate with Primary Children's Hospital (PCH) in Salt Lake City, UT to conduct practical pilot testing of tools and measures refined in Aims 1-3.

The investigators anticipate that knowledge gained from a neonatal safety model developed from data collected prospectively at three children's hospitals and tested within PCH will guide future intervention studies.

A product of the project will be a patient safety registry for surgical neonates. The registry will include a sample of approximately 500 neonatal patients receiving first-time non-cardiac surgical intervention at Monroe Carell Jr. Children's Hospital at Vanderbilt. Neonates who receive NICU care both pre- and post-operatively will be eligible for this study. The registry will include the following data elements: NRE data captured prospectively in the NICU pre-operatively, intraoperatively, and post-operatively, respectively, by trained observers; contributory factors including factors related to patients, clinicians, equipment, logistics, and work environment; and 30-day National Surgical Quality Improvement Project-Pediatric (NSQIP-P) morbidity and mortality outcomes. NRE severity will be categorized and coded as:

1. Serious Safety Event (SSE);
2. Precursor Safety Event (PSE), or
3. Near Miss Safety Event (NME) based on the Safety Event Classification (SEC) system taxonomy.

Surgical morbidity will be categorized using the NSQIP-P taxonomy and classified as Serious (Moderate Temporary Harm to Severe Permanent Harm) or Not Serious (No Harm to Minimal Permanent Harm) using the SEC definitions of levels of harm.

ELIGIBILITY:
Inclusion Criteria:

* Surgical neonates
* Pre- and post-operative care provided in the NICU

Exclusion Criteria:

* neonates having cardiac surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonates undergoing first-time non-cardiac surgeries and who are treated in the neonatal intensive care unit both pre-operatively and post-operatively.
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2016-11; Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
National Surgical Quality Improvement Pediatric Mortality | 30-day
  American College of Surgeons (ACS) NSQIP Pediatric is a nationally validated, risk-adjusted, outcomes-based approach to measure and improve the quality of surgical care for pediatric patients. It employs a prospective, peer-controlled, validated database to quantify 30-day, risk-adjusted surgical outcomes, which provide a valid comparison of outcomes among all hospitals in the program.

SECONDARY OUTCOMES:
National Surgical Quality Improvement Pediatric Morbidity | 30-day
  American College of Surgeons (ACS) NSQIP Pediatric is a nationally validated, risk-adjusted, outcomes-based approach to measure and improve the quality of surgical care for pediatric patients. It employs a prospective, peer-controlled, validated database to quantify 30-day, risk-adjusted surgical outcomes, which provide a valid comparison of outcomes among all hospitals in the program.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J France, PhD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Only aggregate de-identified data will be disseminated.